CLINICAL TRIAL: NCT04777786
Title: Implementation of a Prospective Surveillance Rehabilitation Model for Women With Breast Cancer - A Randomized Controlled Trial
Brief Title: Early Rehabilitation for Breast Cancer - A Randomized Control Trial
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of enrolled participants
Sponsor: University of South Carolina (Other)
Collaborators: Prisma Health-Midlands (Other)
Responsible Party: Principal Investigator, Shana Harrington, Clinical Associate Professor, University of South Carolina
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 115300-20-52703
Record Dates: First submitted 2021-02-16; First posted 2021-03-02 (Actual); Last update posted 2023-11-30 (Actual); Status verified 2023-11

CONDITIONS: Neoplasms, Breast
MeSH Terms: conditions — Breast Neoplasms | interventions — Physical Therapy Modalities

STUDY DESIGN:
Intervention Model Description: Randomized clinical trial design
Who Masked: Outcomes Assessor
Masking Description: Outcomes assessors will be blinded to participant group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Physical Therapy Intervention (Experimental): Individualized physical therapy treatments will be provided based on impairments identified during assessments. Treatment may include but is not limited to the following: passive, assisted and active ROM, manual therapy, soft tissue massage, myofascial release, therapeutic activities and exercise and patient education. Treatment duration and frequency will be specific to each patient, providing personalized care. This type of intervention is considered a pragmatic approach, which will allow for generalization of the results due to the similarity with clinical practice.71 Pilot data indicates women will receive physical therapy intervention 1-2x/week for 3-6 weeks beginning ~4 weeks after surgery (x̄=10 visits).
  Interventions: Other: Physical Therapy
- Usual Care (No Intervention): The usual care group will be instructed to continue with their typical daily activities.

INTERVENTIONS:
Other: Physical Therapy — Individualized physical therapy treatments will be provided based on impairments identified during assessments. Treatment may include but is not limited to the following: passive, assisted and active ROM, manual therapy, soft tissue massage, myofascial release, therapeutic activities and exercise and patient education. Treatment duration and frequency will be specific to each patient, providing personalized care. This type of intervention is considered a pragmatic approach, which will allow for generalization of the results due to the similarity with clinical practice.71 Pilot data indicates women will receive physical therapy intervention 1-2x/week for 3-6 weeks beginning ~4 weeks after surgery (x̄=10 visits).
  Arms: Physical Therapy Intervention

SUMMARY:
Upper extremity strength, range of motion, activity limitations, fatigue and pain are well-documented concerns for women receiving treatment for breast cancer. Research has shown that cancer-related treatment side effects are amenable to rehabilitation interventions when identified early during treatment for breast cancer. Despite this, early rehabilitation has been reported in only 1-2% of individuals diagnosed with cancer. The Prospective Surveillance Model (PSM), a comprehensive model of survivorship care supported by the American Cancer Society and the National Cancer Institute, recommends a baseline assessment (near the time of diagnosis) and ongoing surveillance and intervention of impairments that minimize the impact of cancer treatments. A significant gap in knowledge currently exists with regards to the effectiveness of employing the PSM.

The purpose of this study is to examine the impact of implementing the PSM on impairments and functional limitations in women diagnosed with breast cancer during the first six months of treatment. A randomized controlled trial will be applied to examine a total of 28 women diagnosed with stage I-III breast cancer who will receive a mastectomy at Prisma Health in Columbia, S.C. Women will be randomized to one of two groups: PSM or usual care.

DETAILED DESCRIPTION:
The overall objective of this study is to examine the impact of employing early rehabilitation by implementing a randomized controlled trial at Prisma Health Midlands on women diagnosed with stage I-III breast cancer who will receive a mastectomy.

The following outcomes will be collected at 3-time points (baseline, 3 months and 6 months post-surgery)

* Objective measures: Upper extremity active range of motion, upper extremity, strength, physical function, and arm volume
* Patient reported (questionnaire) measures: Upper extremity function, functional mobility, balance, health-related quality f life, pain, fatigue, falls and distress.

The patient reported measures will also be collected electronically 24 hours after each of the 3 assessments (baseline, 3 months and 6 months post-surgery)

Each of the 3 study visits will last ~60 minutes.

If you are randomized into the intervention group, you will receive ~10 treatment visits with a licensed physical therapist. Scheduling will be at your convenience and based on what the physical therapist recommends. Those in the intervention group will receive individualized physical therapy treatments based on impairments identified. Treatment may include but is not limited to the following: passive, assisted and active ROM, manual therapy, soft tissue massage, myofascial release, therapeutic activities and exercise and patient education. Treatment duration and frequency will be specific to each patient, providing personalized care. Physical therapy intervention will occur 1-2x/week for 3-6 weeks beginning ~4 weeks after surgery (x̄=10 visits). Each visit will last ~60 minutes in duration.

The usual care groups will be instructed to continue with their typical daily activities.

All study participants will receive a handout containing education and home exercise instruction which is considered routine care.

Participants will receive a $25 gift card gift card for each completed in person assessment (baseline, 3 and 6 months post surgery) for a total of $75.

ELIGIBILITY:
Inclusion Criteria:

* Eligible participants include adult female patients, ≥18 years of age, with a primary first-time diagnosis of breast cancer, and referred on or after January 1, 2021 for mastectomy surgery.

Exclusion Criteria:

* Women will be excluded if they will have bilateral surgery, breast-conserving surgery, recurrence of breast cancer, stage IV, or neoadjuvant treatment prior to surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Females with breast cancer are the population of interest.
Enrollment: 3 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2023-03-31 (Actual)

PRIMARY OUTCOMES:
Change in Active range of motion | Pre-surgery (baseline), 3- and 6-months post-surgery.
  Active range of motion (AROM) will be measured in degrees. Measures will include shoulder flexion, external rotation at 90° of shoulder abduction, and shoulder abduction

SECONDARY OUTCOMES:
Upper extremity strength | Pre-surgery (baseline), 3- and 6-months post-surgery.
  Bilateral peak muscle force in pounds will be assessed for shoulder internal rotation, shoulder external rotation, shoulder scaption, and shoulder horizontal adduction.
Upper Extremity Function | Pre-surgery (baseline), 3- and 6-months post-surgery.
  Patient-Reported Outcomes Measurement Information System (PROMIS) Bank v2.0 - Physical Function will be used to assess Upper Extremity Function. Patient-Reported Outcomes Measurement Information System (PROMIS) Bank v2.0 - Physical Function is a computer adaptive test (CAT) where items related to physical function are dynamically selected for administration from an item bank based on the respondent's previous answers. Usually 4-12 items are answered with a high level of measurement precision.
Upper Extremity Function | Pre-surgery (baseline), 3- and 6-months post-surgery.
  The Disabilities of Arm, Shoulder and Hand (DASH) will be used to assess Upper Extremity Function. The Disabilities of Arm, Shoulder and Hand is a 30-item questionnaire designed to assess patient-reported upper limb function. Scores range from 0-100, with higher scores indicating greater disability.
Balance | Pre-surgery (baseline), 3- and 6-months post-surgery.
  Problems with balance will be determined based on the following question: "In the past 12 months (or since the last visit), have you had a problem with balance or difficulty walking? 1 = Yes, 2 = No".
Health-Related Quality of Life | Pre-surgery (baseline), 3- and 6-months post-surgery. 24 hours after baseline assessment, 24 hours after 3-and 6-month post-surgery assessments
  The Functional Assessment of Cancer Therapy-Breast version 4 will assess Health-Related Quality of Life. The Functional Assessment of Cancer Therapy-Breast version 4 is a self-report measure and consists of six domains: physical well-being, social/family well-being, emotional well-being, functional well-being, relationship with doctor, and additional concerns that encompass 41 questions. The higher the score, the better the QOL. Total Functional Assessment of Cancer Therapy-Breast+4 total score ranges 0-148, physical well-being subscale scores range 0-28, social/family well-being subscale scores range 0-28, emotional well-being subscale scores range 0-24, functional well-being subscale scores range 0-28, breast cancer subscale subscale scores range 0-40, arm subscale scores range 0-20.
NCCN Distress Thermometer | Pre-surgery (baseline), 3- and 6-months post-surgery. 24 hours after baseline assessment, 24 hours after 3-and 6-month post-surgery assessments
  The NCCN distress thermometer is a brief screening tool that assesses distress in individuals diagnosed with cancer. This is a patient report measure with an 11-point scale from 0 (no distress) to 10 (extreme distress)
NCCN Distress Problem list | Pre-surgery (baseline), 3- and 6-months post-surgery. 24 hours after baseline assessment, 24 hours after 3-and 6-month post-surgery assessments
  The NCCN distress problem list is a brief screening tool that assesses distress in individuals diagnosed with cancer. The problem checklist is answered yes or no and asks whether the indicated level of distress is related to practical, family, emotional, spiritual/religious, or physical problems
Pain interference | Pre-surgery (baseline), 3- and 6-months post-surgery. 24 hours after baseline assessment, 24 hours after 3-and 6-month post-surgery assessments
  Pain will be measured using the Patient-Reported Outcomes Measurement Information System (PROMIS) Bank v1.1 - Pain interference scale. This is a computer adapted test (CAT) where items related to pain interference are dynamically selected for administration from an item bank based on the respondent's previous answers. Usually 4-12 items are answered for each tool with a high level of measurement precision
Pain intensity | Pre-surgery (baseline), 3- and 6-months post-surgery. 24 hours after baseline assessment, 24 hours after 3-and 6-month post-surgery assessments
  Pain intensity will be measured using the Patient-Reported Outcomes Measurement Information System (PROMIS) Scale v1.0 - Pain intensity 3a. This is a computer adapted test (CAT) where items related to pain intensity are dynamically selected for administration from an item bank based on the respondent's previous answers. Usually 4-12 items are answered for each tool with a high level of measurement precision
Fatigue | Pre-surgery (baseline), 3- and 6-months post-surgery. 24 hours after baseline assessment, 24 hours after 3-and 6-month post-surgery assessments
  Fatigue will be assessed using the 10-point numeric rating scale (NRS) for fatigue and the PROMIS Bank v1.0 Fatigue
Falls | Pre-surgery (baseline), 3- and 6-months post-surgery.
  Falls in the past 12 months (or since the last visit) will be determined by the following question: "Did you fall in the past 12 months (or since the last visit)? 1 = Yes, 2 = No".
Arm volume | Pre-surgery (baseline), 3- and 6-months post-surgery.
  Arm volume will be assessed by taking circumferential measures using a standard 8mm wide flexible tape measure which will then be used to calculate limb volume using a frustum cone.
2-minute step test | Pre-surgery (baseline), 3- and 6-months post-surgery.
  To perform the 2-minute step test, the participant will stand next to a wall, without touching, and march in place raising the knees to a marked target on the wall. This target is midway between the lateral epicondyle of the femur, or the lower thigh bone, and the ASIS or the prominent hip bone. The number of times the right knee reaches the marked target over a 2-minute period will be recorded
30 second sit to stand | Pre-surgery (baseline), 3- and 6-months post-surgery.
  The 30 second sit to stand will be administered using an 18-inch standard office chair without wheels. Starting in a seated position, the patient will fold their arms across their chest without using the armrests or assistance and perform as many sit to stand repetitions as possible in 30 seconds.
Timed arm curl | Pre-surgery (baseline), 3- and 6-months post-surgery.
  , a 5lb weight will be used perform a bicep curl in a seated position. For the starting position, the palm should be facing the participant's body in a resting position. The arm should then rotate so the palm of their hand faces the shoulder at the end of the arm curl. The number of arm curls will be recorded. This will be done on each side.
Timed up and go | Pre-surgery (baseline), 3- and 6-months post-surgery.
  The timed up and go will be administered in a ten-foot walking path marked by a cone. The participant will start in a seated position in a standard office chair without wheels. Time is recorded in seconds while they stand up, walk around the cone and return to a seated position.

CONTACTS AND LOCATIONS:
Locations (1):
- University of South Carolina, Columbia, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Harrington S, Padua D, Battaglini C, Michener LA, Giuliani C, Myers J, Groff D. Comparison of shoulder flexibility, strength, and function between breast cancer survivors and healthy participants. J Cancer Surviv. 2011 Jun;5(2):167-74. doi: 10.1007/s11764-010-0168-0. Epub 2011 Jan 12. PMID 21225372
- [Background] Becker, A.M., Vanlandingham, S., Grogan, M.M., McGowan, M.H., Harrington, S.E. (2019) Impact of Early Rehabilitation in Women Actively Receiving Treatment for Breast Cancer. Rehabilitation Oncology. 38(1): E20, January 2020.
- [Background] Harrington SE, Stout NL, Hile E, Fisher MI, Eden M, Marchese V, Pfalzer LA. Cancer Rehabilitation Publications (2008-2018) With a Focus on Physical Function: A Scoping Review. Phys Ther. 2020 Mar 10;100(3):363-415. doi: 10.1093/ptj/pzz184. PMID 32043151
- [Background] Stout NL, Binkley JM, Schmitz KH, Andrews K, Hayes SC, Campbell KL, McNeely ML, Soballe PW, Berger AM, Cheville AL, Fabian C, Gerber LH, Harris SR, Johansson K, Pusic AL, Prosnitz RG, Smith RA. A prospective surveillance model for rehabilitation for women with breast cancer. Cancer. 2012 Apr 15;118(8 Suppl):2191-200. doi: 10.1002/cncr.27476. PMID 22488693
- [Background] Stout NL, Silver JK, Raj VS, Rowland J, Gerber L, Cheville A, Ness KK, Radomski M, Nitkin R, Stubblefield MD, Morris GS, Acevedo A, Brandon Z, Braveman B, Cunningham S, Gilchrist L, Jones L, Padgett L, Wolf T, Winters-Stone K, Campbell G, Hendricks J, Perkin K, Chan L. Toward a National Initiative in Cancer Rehabilitation: Recommendations From a Subject Matter Expert Group. Arch Phys Med Rehabil. 2016 Nov;97(11):2006-2015. doi: 10.1016/j.apmr.2016.05.002. Epub 2016 May 27. PMID 27237580
- [Background] Schmitz KH, Stout NL, Andrews K, Binkley JM, Smith RA. Prospective evaluation of physical rehabilitation needs in breast cancer survivors: a call to action. Cancer. 2012 Apr 15;118(8 Suppl):2187-90. doi: 10.1002/cncr.27471. No abstract available. PMID 22488692
- [Background] Stout NL, Andrews K, Binkley JM, Schmitz KH, Smith RA. Stakeholder perspectives on dissemination and implementation of a prospective surveillance model of rehabilitation for breast cancer treatment. Cancer. 2012 Apr 15;118(8 Suppl):2331-4. doi: 10.1002/cncr.27470. PMID 22488707